CLINICAL TRIAL: NCT00893165
Title: Does Moderate Physical Activity in Chronic Hemodialysis Patients Reduce Inflammation Via Inhibition of Proinflammatory Monocyte Activity?
Brief Title: Does Moderate Physical Activity in Hemodialysis Patients Reduce Inflammation?
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Matthias Girndt, Professor of Internal Medicine, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: KIM2H-2009-01; Roux 19/39; KfH 2009-0010
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: End-stage Renal Disease; Hemodialysis
Keywords: inflammation; cardiovascular disease
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and DNA samples

GROUPS / COHORTS (1):
- hemodialysis patients: chronic hemodialysis patients with elevated inflammation markers
  Interventions: Behavioral: moderate physical activity

INTERVENTIONS:
Behavioral: moderate physical activity — bed mounted cycles for physical activity for 30 min during each hemodialysis session

SUMMARY:
The purpose of this study is to observe a potential benefit of moderate physical activity by using bed mounted cycles during hemodialysis treatment sessions on inflammatory markers in the blood of patients with end-stage renal disease (ESRD).

DETAILED DESCRIPTION:
Patients with ESRD on chronic hemodialysis patients frequently have elevated markers of inflammation (e.g., serum CRP values) and accumulation of proinflammatory monocyte populations in the circulation. The level of inflammation is highly predictive for cardiovascular disease and mortality. Physical activity has been shown to improve dialysis efficacy by improving the elimination of retention solutes. In healthy individuals, sports activity influences inflammatory immune parameters. The study will observe the influence of moderate physical activity (using a bed mounted cycle for 30min during dialysis thrice weekly) on circulating monocyte subpopulations and inflammatory proteins over a 9 month period in 16 chronic hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis treatment for at least three months
* three dialysis sessions per week
* good general clinical condition
* stable hemodynamics during the most recent three dialysis sessions

Exclusion Criteria:

* conditions making the patient unable to use the bed mounted cycle (amputations, joint disease etc)
* clinically obvious acute infections
* active malignancy
* pathologic results of spiroergometry or echocardiography that imply an elevated risk of participation
* myocardial infarction within the last 12 weeks
* uncontrolled arterial hypertension
* uncontrolled diabetes mellitis with frequent hypoglycemia
* unability to understand and consent the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients on chronic hemodialysis therapy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Composition of monocyte subpopulations as defined by CD14 and CD16 expression | 6 months

SECONDARY OUTCOMES:
Serum CRP values | 6 months
Dialysis quality (kt/V, URR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Girndt, MD, Study Director — Martin-Luther-University Halle-Wittenberg, Germany
Locations (1):
- Department of Internal Medicine II, Halle, Saxony-Anhalt, Germany